CLINICAL TRIAL: NCT02040324
Title: Comparison of Lung Function in Patients After Lower Abdominal Surgery Exceeding 2hrs Under the Use of Laryngeal Mask vs. Endotracheal Tube for Airway Management
Brief Title: Laryngeal Mask Airway in Lower Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Daniel Reuter, Professor of Anesthesiology, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LMA UKE
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Major Lower Abdominal Surgery
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotracheal Intubation (Active Comparator): Clinical routine for longer lasting procedures
  Interventions: Device: Endotracheal tube
- Laryngeal Mask (Experimental): Laryngeal mask with gastric access and drainage as airway management instead of endotracheal intubation
  Interventions: Device: Laryngeal mask with gastric access

INTERVENTIONS:
Device: Laryngeal mask with gastric access
  Arms: Laryngeal Mask
Device: Endotracheal tube
  Arms: Endotracheal Intubation

SUMMARY:
We measure in this study lung function of 100 patients immediately after major lower abdominal surgery. We compare lung function, when either endotracheal intubation, or laryngeal masks are used for airway protection during surgery. The hypothesis is that the use of laryngeal masks is associated with less impairment of lung function in the immediate postoperative phase.

ELIGIBILITY:
Inclusion Criteria - patients scheduled for elective retropubic radical prostatectomy

Exclusion Criteria:

- increased risk of aspiration due to hiatal hernia, morbid obesity, or facial malformations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The change between pre- and postoperative forced expiratory volume in one second (FEV1) in lung function | one day prior to surgery, 1 hour after surgery (recovery room), at day one after surgery
  The lung function is quantified by using Spirometry and pulse oximetry. Spirometry is performed in a standardized way according to the recommendations of the American Thoracic Society (ATS) and European Respiratory Society (ERS)

SECONDARY OUTCOMES:
Vital capacity (VC) measured by spirometry. | one day prior to surgery, i hour after after surgery (recovery room), at day one after surgery
  Spirometry is performed in a standardized way according to the recommendations of the American Thoracic Society (ATS) and European Respiratory Society (ERS)
Forced vital capacity (FVC) | one day prior to surgery, one hour after surgery (recovery room), at day one after surgery
mid-expiratory flow (MEF 25, 50, 75) | one day prior to surgery, one hour after surgery, at day one after surgery
Peak expiratory flow (PEF) | one day prior to surgery, one hour after surgery (recovery room) , at day one after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Reuter, MD, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf